CLINICAL TRIAL: NCT04022161
Title: Effects of Prolonged Delivery of Nitric Oxide Gas on Plasma Reduction-Oxidation Reactions in Cardiac Surgical Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Zadek, Francesco, M.D., Massachusetts General Hospital (Unknown); Spina, Stefano, M.D., Massachusetts General Hospital (Unknown); Marrazzo, Francesco, M.D., Massachusetts General Hospital (Unknown); University of Southampton (Other)
Responsible Party: Principal Investigator, Lorenzo Berra, MD, Lorenzo Berra, MD, Associate Professor of Anesthesia, Critical Care and Pain Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: RedOx-NO
Record Dates: First submitted 2019-07-10; First posted 2019-07-16 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cardiovascular Diseases; Oxidative Stress; Endothelial Dysfunction
Keywords: Cardiac surgery; Nitric oxide; Oxidative Stress; Redox Thiols couples; Lipids peroxidation; Protein Oxidation
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Nitrogen; Inhalation; Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrogen (Placebo Comparator): Inhaled nitrogen will be administered via the cardiopulmonary bypass (CPB) machine and after CPB via the inspiratory limb of the anesthetic or ventilator circuit, and thereafter via the mechanical ventilator in the Intensive Care Unit (ICU). Test gas administration will commence at the onset of CPB and last for 24 hours.
  Interventions: Drug: Nitrogen Gas for Inhalation; Other: Blood withdrawal
- Nitric Oxide (Experimental): Inhaled nitric oxide (iNO) will be administered via the cardiopulmonary bypass (CPB) machine and after CPB via the inspiratory limb of the anesthetic or ventilator circuit, and thereafter via the mechanical ventilator in the ICU. Test gas administration will commence at the onset of CPB and last for 24 hours. At the end of 24 hours, inhaled nitric oxide (iNO) will be weaned and discontinued.
  Interventions: Other: Blood withdrawal; Drug: Nitric Oxide

INTERVENTIONS:
Drug: Nitrogen Gas for Inhalation — See arm description
  Other Names: N2
  Arms: Nitrogen
Other: Blood withdrawal — Blood samples will be collected over four time-points: (I) baseline (before surgery) (II) end of the surgery, (III) end of 24 hours of gas delivery and (IV) 24 hours from the gas suspension.
Drug: Nitric Oxide — See arm description
  Other Names: iNO
  Arms: Nitric Oxide

SUMMARY:
This study is an ancillary (add-on) study to the clinical trial entitled "Effect of Nitric Oxide in Cardiac Surgery Patients With Endothelial Dysfunction", which has Clinical Trials.gov identifier NCT02836899. NCT02836899 trial randomizes cardiac surgical patients to receive either Nitric Oxide (NO) or a placebo during and after cardiac surgery.

This ancillary study aims to assess the effects of Nitric Oxide on plasma reduction-oxidation reactions of patients undergoing cardiac surgery requiring prolonged cardiopulmonary bypass.

DETAILED DESCRIPTION:
The endothelial dysfunction is a pathologic process characterized by impaired endothelial nitric oxide (NO) signaling and metabolism leading to decreased vascular response to vasodilation. Cardiac surgical patients affected by multiple cardiovascular risk factors (e.g., hypertension, diabetes, dyslipidemia) commonly present with endothelial dysfunction due to a chronic unbalance of the redox state caused by an increased oxidative stress. Moreover, the use of cardiopulmonary bypass, the hemolysis, the ischemia and the inflammation associated with the surgery magnifies the oxidative stress, which has been shown to contribute to post-operative complications. In order to decrease oxidative stress, several antioxidant drugs and vitamins have been trialed with marginal health benefits.

Recently, different research groups reported that NO delivered during cardiac surgery improved outcomes both in children and adults. Nitric oxide decreased the incidence and the severity of postoperative acute kidney injury, the extension of infarction size, the duration of mechanical ventilation, the length of stay and the use of rescue therapies as postoperative venous-arterial extra-corporeal membrane oxygenation.

The exogenous administration of NO has been shown to prevent the scavenging of endogenous NO by inactivating the highly oxidative-reactive ferrous plasma oxy-hemoglobin to ferric met-hemoglobin. Our group is conducting a randomized controlled trial at Massachusetts General Hospital (Boston, USA) in patients with signs and symptoms of endothelial dysfunction, undergoing cardiac surgery requiring prolonged cardiopulmonary bypass and randomized to receive NO or placebo. However, the mechanisms underlying the effects of NO admistration on plasmatic redox equilibrium have still to be determined. The aim of this ancillary study is (I) to determine the changes of redox state in the plasma of surgical patients receiving either 80 ppm of NO (study group) or Nitrogen (placebo group). (II) To evaluate whether the degree of change in redox state is associated to postoperative complication.

ELIGIBILITY:
Inclusion Criteria:

* Eligible and randomized in the trial NCT02836899
* Provide written informed consent
* Age ≥ 18 years of age
* Elective cardiac or aortic surgery with CPB >90 minutes
* Clinical evidence of endothelial dysfunction assessed by a specifically designed questionnaire

Exclusion Criteria:

* Estimated Glomerular Filtration Rate less than 30 ml/min/1.73 m2
* Emergent cardiac surgery
* Life expectancy < 1 year at the time of enrollment
* Hemodynamic instability as defined by a systolic blood pressure <90 mmHg.
* Mean pulmonary artery pressure ≥ 40 mm Hg and PVR > 4 Wood Units.
* Left ventricular ejection fraction < 30% by echocardiography obtained within three months of enrollment
* Administration of one or more Packed Red Blood Cell (PRBC) transfusions in the week prior to enrollment
* X-ray contrast infusion less than 48 hours before surgery
* Evidence of hemolysis from any other origin:

  a. Intravascular: i. Intrinsic RBC defects leading to hemolytic anemia (eg, enzyme deficiencies, hemoglobinopathies, membrane defects) ii. Extrinsic: liver disease, hypersplenism, infections (eg, bartonella, babesia, malaria), treatment with oxidizing exogenous agents (eg, dapsone, nitrites, aniline dyes), exposure to other hemolytic agents (eg, lead, snake and spider bites), lymphocyte leukemia, autoimmune hemolytic disorders b. Extravascular: Infection (eg, clostridial sepsis, severe malaria), paroxysmal cold hemoglobinuria, cold agglutinin disease, paroxysmal nocturnal hemoglobinuria, iv infusion of Rho(D) immune globulin, iv infusion of hypotonic solutions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2025-11-24 (Actual); Study Completion 2025-11-24 (Actual)

PRIMARY OUTCOMES:
Changes in the concentration of glutathione/glutathione disulfide (GSH/GSSG) and the cysteine/ cysteine disulfide (Cys/CysSS) couples in the plasma after cardiac surgery. | Plasma will be sampled before the cardiac surgery and during the first 48 hours from surgery
  The investigators will measure the changes in plasma concentration of GSH, GSSG, Cys, CysSS, of subjects undergoing cardiac surgery with prolonged cardiopulmonary bypass, using ultrahigh-performance liquid chromatography in combination with electrospray-ionization tandem mass spectrometry. The concentration will be expressed in microMoles.
Changes in the electrical potential of glutathione/glutathione disulfide (GSH/GSSG) and the cysteine/ cysteine disulfide (Cys/CysSS) couples in the plasma after cardiac surgery. | Plasma will be sampled before the cardiac surgery and during the first 48 hours from surgery
  The investigators will compare the changes of plasma redox state from baseline of patients receiving either 80 ppm of nitric oxide (study group) or nitrogen (placebo group), during cardiac surgery. The redox state will be assessed by measuring the electrical potential of GSH/GSSG and the Cys/CysSS couples in the plasma, using Nerst's equation. The electrical potential will be express in milliVolt.

SECONDARY OUTCOMES:
Changes of concentration in plasma and red blood cells of nitric oxide metabolites after cardiac surgery. | Plasma will be sampled before the cardiac surgery and after the first 48 hours from surgery
  The investigators will describe the trends in plasma and red blood cells of nitric oxide (NO) metabolites after the surgery. Nitric oxide (NO) metabolites concentrations will be measured using chemiluminescence. The concentrations will be expressed in microMoles.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Berra, MD, Principal Investigator — Massachusett General Hospital
Locations (2):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- MP 825 Southampton General Hospita, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marrazzo F, Spina S, Zadek F, Lama T, Xu C, Larson G, Rezoagli E, Malhotra R, Zheng H, Bittner EA, Shelton K, Melnitchouk S, Roy N, Sundt TM, Riley WD, Williams P, Fisher D, Kacmarek RM, Thompson TB, Bonventre J, Zapol W, Ichinose F, Berra L. Protocol of a randomised controlled trial in cardiac surgical patients with endothelial dysfunction aimed to prevent postoperative acute kidney injury by administering nitric oxide gas. BMJ Open. 2019 Jul 4;9(7):e026848. doi: 10.1136/bmjopen-2018-026848. PMID 31278097
- [Background] Sutton TR, Minnion M, Barbarino F, Koster G, Fernandez BO, Cumpstey AF, Wischmann P, Madhani M, Frenneaux MP, Postle AD, Cortese-Krott MM, Feelisch M. A robust and versatile mass spectrometry platform for comprehensive assessment of the thiol redox metabolome. Redox Biol. 2018 Jun;16:359-380. doi: 10.1016/j.redox.2018.02.012. Epub 2018 Feb 19. PMID 29627744